CLINICAL TRIAL: NCT04579822
Title: Maternal and Fetal Outcomes Following Influenza Vaccination in Pregnancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sungkyunkwan University (Other)
Collaborators: Government-wide R&D Fund project for infectious disease research (GFID) (Unknown)
Responsible Party: Principal Investigator, Ju-Young Shin, Associate Professor, Sungkyunkwan University
Other Study IDs: SKKU-2020-FP
Record Dates: First submitted 2020-09-28; First posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy Related; Influenza Virus Vaccine Adverse Reaction
MeSH Terms: interventions — Influenza Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women vaccinated with a QIV: Women aged 20-44 years who had received a QIV during their pregnancy between September 22, 2020, and April 30, 2021, under the national immunization program in South Korea.
  Interventions: Biological: influenza vaccine
- Pregnant women unvaccinated with a QIV: Women aged 20-44 years who had not received a QIV during their pregnancy between September 22, 2020, and April 30, 2021, under the national immunization program in South Korea.
  Interventions: Biological: influenza vaccine

INTERVENTIONS:
Biological: influenza vaccine — quadrivalent influenza vaccination in the flu seasons

SUMMARY:
This is a nationwide cohort study to assess maternal and fetal outcomes following vaccination with a quadrivalent influenza vaccine (QIV) during pregnancy.

DETAILED DESCRIPTION:
The Korean National Immunization Program (NIP) first introduced quadrivalent influenza immunization for all pregnant women in the 2020-2021 season. This nationwide cohort study is proposed to assess the risks of adverse maternal and fetal outcomes following vaccination with a quadrivalent influenza vaccine (QIV) during pregnancy. We will use the national health insurance database from the National Health Insurance Service (NHIS) linked with the national immunization program registry data from the Korea Centers for Diseases Control & Prevention (KCDC).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between September 22, 2020, and April 30, 2021.

Exclusion Criteria:

* Women aged <20 or >45 years
* Pregnancies with a chromosomal abnormality
* Pregnancies with exposure to a known teratogenic medication

Ages: 20 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women during the period of the national immunization program in South Korea.
Sampling Method: Probability Sample
Enrollment: 300000 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-10-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk of adverse pregnancy outcomes | from delivery up to 1 year after birth
  Spontaneous abortion, stillbirth, neonatal death, congenital anomaly, pre-term birth, fetal growth restriction, small for gestational age, and low birth weight, which are confirmed by diagnostic records in the NHIS database.
Risk of vaccine-related adverse events | from delivery up to 1 year after birth
  Vaccine-related adverse events confirmed by diagnostic records in the NHIS database.
Risk of poor health outcomes in pregnant women | from delivery up to 1 year after birth
  Hospital admission, emergency department visits, influenza infection, and hospitalization with influenza infection, which are confirmed by diagnosis and healthcare utilization records in the NHIS database.
Risk of poor health outcomes in neonates | from delivery up to 1 year after birth
  Respiratory distress, neonatal intensive care unit admission, and hospital visits with neonatal infection or fever, which are confirmed by diagnosis and healthcare utilization records in the NHIS database.

SECONDARY OUTCOMES:
Risk of pregnancy-related complications | from delivery up to 1 year after birth
  Pre-eclampsia/eclampsia, gestational diabetes mellitus, antenatal bleeding, postpartum hemorrhage, and maternal death, which are confirmed by diagnostic records in the NHIS database.

CONTACTS AND LOCATIONS:
Overall Officials: Ju-Young Shin, PhD, Principal Investigator — Sungkyunkwan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baum U, Leino T, Gissler M, Kilpi T, Jokinen J. Perinatal survival and health after maternal influenza A(H1N1)pdm09 vaccination: A cohort study of pregnancies stratified by trimester of vaccination. Vaccine. 2015 Sep 11;33(38):4850-7. doi: 10.1016/j.vaccine.2015.07.061. Epub 2015 Aug 1. PMID 26238723
- [Background] Macias Saint-Gerons D, Sola Arnau I, De Mucio B, Arevalo-Rodriguez I, Aleman A, Castro JL, Ropero Alvarez AM. Adverse events associated with the use of recommended vaccines during pregnancy: An overview of systematic reviews. Vaccine. 2021 Jul 30;39 Suppl 2:B12-B26. doi: 10.1016/j.vaccine.2020.07.048. Epub 2020 Sep 21. PMID 32972737
- [Background] Walsh LK, Donelle J, Dodds L, Hawken S, Wilson K, Benchimol EI, Chakraborty P, Guttmann A, Kwong JC, MacDonald NE, Ortiz JR, Sprague AE, Top KA, Walker MC, Wen SW, Fell DB. Health outcomes of young children born to mothers who received 2009 pandemic H1N1 influenza vaccination during pregnancy: retrospective cohort study. BMJ. 2019 Jul 10;366:l4151. doi: 10.1136/bmj.l4151. PMID 31292120
- [Background] Ludvigsson JF, Strom P, Lundholm C, Cnattingius S, Ekbom A, Ortqvist A, Feltelius N, Granath F, Stephansson O. Maternal vaccination against H1N1 influenza and offspring mortality: population based cohort study and sibling design. BMJ. 2015 Nov 16;351:h5585. doi: 10.1136/bmj.h5585. PMID 26572546
- [Background] Hviid A, Svanstrom H, Molgaard-Nielsen D, Lambach P. Association Between Pandemic Influenza A(H1N1) Vaccination in Pregnancy and Early Childhood Morbidity in Offspring. JAMA Pediatr. 2017 Mar 1;171(3):239-248. doi: 10.1001/jamapediatrics.2016.4023. PMID 27893898